CLINICAL TRIAL: NCT05546788
Title: The Effectiveness of Hydroxylated Polymethoxy Flavones Solid Dispersion Incorporated Sodium Carboxymethyl Cellulose Gel With Periodontal Debridement in the Treatment of Periodontitis. Clinical- Biochemical Study
Brief Title: Hydroxylated Polymethoxy Flavones Solid Dispersion in Treatment of Periodontitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mortada, Head of Department of Oral Medicine, Periodontology and Diagnosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.S.V.U 122/22
Record Dates: First submitted 2022-09-04; First posted 2022-09-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Disease; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Three groups of patients with periodontitis, Group I received plain gel Group II received chlorhexidine gel Group III received hydroxylated polymethoxy flavones solid dispersion gel
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- hydroxylated polymethyl flavones group (Active Comparator): SRP then hydroxylated polymethyl flavones addition
  Interventions: Procedure: scaling and root planing; Drug: hydroxylated poly methoxy flavones
- Chlorohexidine group (Active Comparator): SRP then Chlorohexidine gel application
  Interventions: Procedure: scaling and root planing; Drug: chlorhexidine
- placebo group (Placebo Comparator): SRP then placebo gel application
  Interventions: Procedure: scaling and root planing; Drug: placebo

INTERVENTIONS:
Procedure: scaling and root planing — subgingival Depridement
Drug: hydroxylated poly methoxy flavones — Received hydroxylated poly methoxy flavones extract solid dispersion incorporated into sodium carboxymethylcellulose gel
  Arms: hydroxylated polymethyl flavones group
Drug: chlorhexidine — Received chlorhexidine gel
  Arms: Chlorohexidine group
Drug: placebo — Received placebo gel
  Arms: placebo group

SUMMARY:
Periodontitis is a serious gum infection that damages the soft tissue and, without treatment, can destroy the bone that supports your teeth.

Hydroxylated poly methoxy flavones are a combination of naturally occurring flavonoids extracted from the orange peel and exert anti-inflammatory, antibacterial, and antifungal activity however, this extract is poorly soluble and poorly absorbable. In this work, this extract was formulated as a solid dispersion formulation to enhance its biological activity and then incorporated into a gel base and used in the treatment of periodontitis after clinical debridement.

DETAILED DESCRIPTION:
In the study, there are 3 groups; the first one first one received plain sodium carboxymethylcellulose. Group II received chlorhexidine gel. GroupIII received Hydroxylated poly methoxy flavones solid dispersion incorporated into sodium carboxymethylcellulose gel.

In all groups, there is clinical debridement before injection of gels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periodontitis stage I-II
* free from any systemic disorders.
* no mobility - non-smokers - no parafunctional habits.
* Each patient with minimum three periodontitis sites ( split-mouth study)

Exclusion Criteria:

* Smokers.
* patients with diabetes, and hypertension.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment loss will be quantified in centimeters before and after treatment | One week
  Should be minimized in the group treated with Hydroxylated Polymethoxy Flavones gel than in other groups
Pocket Depth will be quantified in centimeters before and after treatment | One week
  Should be minimized in the group treated with Hydroxylated Polymethoxy Flavones gel

IPD SHARING:
Plan to Share IPD: No